CLINICAL TRIAL: NCT02502032
Title: Effects of Pretreatment With Different Doses of Cisatracurium on Succinylcholine-induced Fasciculations
Brief Title: Effects of Cisatracurium on Sccinylcholine-induced Fasciculations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhuan Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhuan Zhang, MD, Yangzhou No.1 People's Hospital
Organization: Yangzhou No.1 People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ZZ0716
Record Dates: First submitted 2015-07-16; First posted 2015-07-17 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Fasciculations
MeSH Terms: conditions — Fasciculation | interventions — cisatracurium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cisatracurium 0.005 mg/kg (Experimental): The group received pretreatment of cisatracurium 0.005 mg/kg.
  Interventions: Drug: Cisatracurium
- Cisatracurium 0.01 mg/kg (Experimental): The group received pretreatment of cisatracurium 0.01 mg/kg.
  Interventions: Drug: Cisatracurium
- Cisatracurium 0.02 mg/kg (Experimental): The group received pretreatment of cisatracurium 0.02 mg/kg.
  Interventions: Drug: Cisatracurium

INTERVENTIONS:
Drug: Cisatracurium — Different groups received different pretreatments of cisatracurium.
  Other Names: Dose

SUMMARY:
To investigate the effects of different doses of cisatracurium pretreatment on succinylcholine-induced fasciculations.

DETAILED DESCRIPTION:
Ninety patients scheduled for laparoscopic cholecystectomies were equally randomized into three groups to receive pretreatment of 0.005, 0.01, and 0.02 mg/kg cisatracurium, respectively. General anesthesia was induced 3.5 min later, train of four stimulation was monitored 4.5 min later, succinylcholine 1.5 mg/kg was injected 5 min later, and endotracheal intubation was implemented 6.5 min later. The side effects of cisatracurium, intensity of fasciculations, intubating conditions, time and extent to maximal depression of twitch and time for its recovery to 20% of control value, severity of myalgia at 24 h postoperatively, serum potassium before cisatracurium pretreatments, at intubating time, and 5 min after intubation were recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Standards Association (ASA) physical status I or II patients scheduled for elective laparoscopic cholecystectomies with tracheal intubation requiring general anesthesia;
* 20 - 65 years old;
* Without acid-base imbalance and electrolyte disturbance;
* With normal hepatic and renal function.

Exclusion Criteria:

* Patients with the contraindications associated with succinylcholine or cisatracurium;
* Patients taking drugs known to alter the action of neuromuscular blockers;
* Patients with a body mass index exceeding 30

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Presence of fasciculations | After the injection of succinylcholine for 1.5 minutes

SECONDARY OUTCOMES:
Side effects of the pretreatment of cisatracurium | From the time of 3 minutes after the pretreatment of cisatracurium for 0.5 minutes
The time to maximal depression of twitch | From the time of 4.5 minutes after the pretreatment of cisatracurium for two minutes
The extent to maximal depression of twitch | From the time of 4.5 minutes after the pretreatment of cisatracurium for two minutes
The grades of endotracheal intubation | At intubating time
The changes of serum potassium | After entering the operating theater till the anesthesia induction, at intubating, and 5 min after intubation
Myalgia at 24 hours postoperatively | At 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Xin-nong Liu, Professor, Study Director — Yangzhou No. 1 Peoples' Hospital